CLINICAL TRIAL: NCT04744233
Title: Effect of Traditional and Emerging Conservation Technologies on Bioactive Compounds and Their Antioxidant Capacity in Plant Foods
Brief Title: Bioavailability of Carotenoids From Orange Juice in a Cross-over Study in Healthy Subjects.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Ciencia y Tecnología de Alimentos y Nutrición (Other Government)
Collaborators: Comunidad de Madrid (Other); Instituto de Salud Carlos III (Other Government); Puerta de Hierro University Hospital (Other)
Responsible Party: Principal Investigator, Begoña Olmedilla, Research Scientist. Ph.D., Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CAM-HUPH-IF
Record Dates: First submitted 2021-01-27; First posted 2021-02-08 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Biological Availability; Carotenoids; Lutein; Humans

STUDY DESIGN:
Intervention Model Description: Multiple dose cross-over study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Freshly squeezed orange juice (FS) (Active Comparator): Subjects were enrolled to consume 500 mL of orange juice/day during three consecutive 14 days periods separated by 1 - 1.5 month washouts. The orange juice assayed was freshly squeezed (FS). Six subjects consumed FS-orange juice.
  Interventions: Other: Orange juice
- Commercially available low pasteurized orange juice (LP) (Active Comparator): Subjects were enrolled to consume 500 mL of orange juice/day during three consecutive 14 days periods separated by 1 - 1.5 month washouts. The orange juices assayed was commercially available low pasteurized juice (LP). All participants consumed the LP orange juices.
  Interventions: Other: Orange juice
- High-pressure processed orange juice(HPP) (Active Comparator): Subjects were enrolled to consume 500 mL of orange juice/day during three consecutive 14 days periods separated by 1 - 1.5 month washouts. The orange juices assayed was high-pressure processed (HPP). All participants consumed the HPP orange juices.
  Interventions: Other: Orange juice
- Pulsed electric fields treated orange juice (PEF) (Active Comparator): Subjects were enrolled to consume 500 mL of orange juice/day during three consecutive 14 days periods separated by 1 - 1.5 month washouts. The orange juices assayed was those treated with pulsed electric fields (PEF). Six participants consumed the PEF-orange juice.
  Interventions: Other: Orange juice

INTERVENTIONS:
Other: Orange juice — Subjects were enrolled to consume 500 mL of orange juice/day during three consecutive 14 days periods separated by 1 - 1.5 month washouts. The orange juices assayed were: freshly squeezed (FS), commercially available low pasteurized juice (LP) and juices treated by high-pressure processing (HPP) and by pulsed electric fields (PEF). All participants consumed the LP and the HPP orange juices. Six subjects consumed PEF-orange juice and other six consumed the FS-orange juice.

SUMMARY:
Commercially available fruit juices are obtained after applying industrial technologies to preserve and extend the shelf-life by inactivation of microorganism and enzymes. These are traditional thermal treatment (eg. pasteurization, sterilization) that causes losses of nutritional and bioactive compounds, changes physicochemical properties (colour, flavor and texture) and can modify their bioavailabilities. Thus, the traditional thermal processing is being replaced by less intense thermal technologies (e.g. low-temperature pasteurization / refrigerated storage) and non-thermal treatments such as the high-pressure processing (HPP) and the pulsed electric fields (PEF) as an alternative to enhace food safety and shelf-life without compromising organoleptic qualities (retain the flavour, color healthiness of fresh foods) and keeping their health-promoting capacity. The beneficial health effect derived from the orange juice intake is partly related to the bioavailability of their bioactive compounds.

The aim of this study was to assess the effect of the intake of freshly squeezed orange juice (Citrus sinensis L.) and processed orange juice elaborated with different treatments (low pasteurization / refrigerated storage, high-pressure processing, pulsed electric fields) on the main serum carotenoid concentrations in a cross-over study in apparently healthy subjects using multiple dosis.

DETAILED DESCRIPTION:
Methods Twelve healthy subjects (6 men), age 20-32 y, were enrolled in a cross-over study, to consume 500 mL of orange juice/day during 14 days periods. All volunteers consumed the LP and HPP, six consumed PEF or FS-orange juice. Fasted blood was collected at baseline and on days 7 and 14. Carotenoid concentrations in serum and orange juice were analyzed by high performance liquid chromatogry (HPLC).

ELIGIBILITY:
Inclusion Criteria:

* age (20- 32 y)
* body mass index (BMI)
* serum cholesterol and triglycerides concentrations within the normal range
* serum retinol within the range 31 - 70 µg/dL.

Exclusion Criteria:

* vitamin / mineral supplements intake
* regular medication
* pregnancy or lactating
* chronic disease
* smoking habit.

Ages: 20 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2001-10 (Actual); Primary Completion 2002-06 (Actual); Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Assessment of the effect of dairy intake of orange juice elaborated with four different procedures on the serum carotenoid concentrations of healthy adults. | 6 months
  Assessment of the effect of dairy intake of orange juice elaborated with low temperature pasterurization (LP), high-pressure processing (HPP), pulsed electric fields (PEF) and freshly squeezd (FS) on the serum carotenoid concentrations of healthy adults.

CONTACTS AND LOCATIONS:
Overall Officials: Olmedilla-Alonso, Principal Investigator — Instituto de Ciencia y Tecnología de Alimentos y Nutrición
Locations (2):
- Spain (2):
  - Madrid
  - Begoña Olmedilla-Alonso, Madrid